CLINICAL TRIAL: NCT07246941
Title: A Phase I, 2-Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single-ascending Doses of Intrathecally Administered RG6496 in a Randomized, Placebo-controlled, Investigator/Participant-blind Study With an Open-label Extension in Huntington's Disease Gene Expansion Carriers
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RG6496 in Huntington's Disease
Acronym: POINT-HD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP45378; 2025-520631-17-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-19; First posted 2025-11-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part 1: Investigator & participants will be blinded; Part 2: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: RG6496 (Experimental): Participants will receive single dose of RG6496. Participants will be enrolled in planned sequential cohorts associated with ascending dose levels.
  Interventions: Drug: RG6496
- Part 1: Placebo (Placebo Comparator): Participants will receive a single dose of RG6496 matching placebo.
  Interventions: Drug: Placebo
- Part 2: OLE (Experimental): All participants who have completed Part 1 and are eligible for Part 2 will receive one open-label dose of RG6496.
  Interventions: Drug: RG6496

INTERVENTIONS:
Drug: RG6496 — RG6496 will be administered as per the schedule specified in the respective arms.
  Arms: Part 1: RG6496; Part 2: OLE
Drug: Placebo — RG6496 matching placebo will be administered as per the schedule specified in placebo arm.
  Arms: Part 1: Placebo

SUMMARY:
This is a first-in-human (FIH) study of RG6496 that will assess the safety and tolerability of single-ascending doses of RG6496 administered to huntington's disease gene expansion carriers (HDGECs). The study consists of two parts: Part 1 [single-ascending dose] followed by Part 2 [open-label extension (OLE)].

ELIGIBILITY:
Inclusion Criteria:

Part 1

* Confirmation of HDGEC status with cytosine-adenine-guanine (CAG) expansion > 39.
* Confirmation of SNP carrier status of the target SNP
* Independence Scale (IS) score of ≥70, total functional capacity (TFC) ≥10, total motor score (TMS) >6.
* Ability to read the words "red," "blue," and "green" and be fluent in the language of the informed consent form (ICF) and the tests used at the study site.
* Ability to walk unassisted.
* Total body weight > 40 kilogram (kg) and body mass index (BMI) within the range 18-32 kilogram per square meter (kg/m^2) (inclusive) at baseline.
* Ability to undergo and tolerate MRI scans.

Part 2

* Completed the post-dose safety follow-up period in the Part 1 of the study.
* In the opinion of the Investigator, the participant has not experienced a worsening in health that precludes their safe continued participation in the study.

Exclusion Criteria:

Part 1

* Concurrent or planned participation in any interventional clinical study, including current use of an ASO or any HTT-lowering therapy or treatment with investigational therapy within 90 days or 5 drug-elimination half-lives, whichever is longer prior to screening
* Pregnant or breastfeeding, or with the intention of becoming pregnant during the study or within the timeframe in which contraception is required
* Malignancy within 5 years prior to screening
* Planned brain surgery during the study
* Positive HIV test, hepatitis B surface antigen and hepatitis B surface antigen at screening
* Active psychosis, confusional state, or violent behavior, including aggression that could cause harm to self or others, over the 12 weeks prior to screening.
* Current or previous history of a primary independent psychotic disorder.
* Scoliosis or spinal deformity or surgery making IT injection not feasible in an outpatient setting
* History of attempted suicide or suicidal ideation with plan (i.e., active suicidal ideation) that required hospital visit and/or change in level of care within 12 months prior to screening.

Part 2

* Prematurely discontinued from Part 1 for any reason (i.e., before the completion of the postdose safety follow-up period of Part 1).
* Pregnant or breastfeeding, or with the intention of becoming pregnant during the study or within the timeframe in which contraception is required.
* Concurrent or planned participation in any interventional clinical study, including current use of an ASO or any HTT-lowering therapy
* Received any active investigational treatment other than RG6496 during or since completion of Part 1 of the study.
* Had confirmed Dose-Limiting Adverse Event (DLAE)(s) in Part 1 of the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-12-11 (Estimated); Study Completion 2029-03-05 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Adverse Events (AEs) | Up to approximately 24 months
Part 1: Change From Baseline in Neurological Assessment | Up to approximately 24 months
  A neurologic examination including fundoscopy, will be performed by a neurologist or an ophthalmologist depending on local practice. A neurologic examination will include an assessment of mental status, level of consciousness, cranial nerve function, motor function, sensory function, reflexes, gait, and coordination.
Part 1: Percentage of Participants With Suicidal Ideation or Behavior, as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Up to approximately 24 months
  C-SSRS measures 4 constructs as follows: severity of ideation, intensity of ideation, behavior, and lethality of actual suicide attempts. Binary (yes/no) data are collected for 10 categories. Numeric ratings are provided for intensity of ideation (if present), from 1 to 5, with 1 being the least severe and 5 being the most severe.
Part 1: Change from Baseline in Montreal Cognitive Assessment (MoCA) | Up to approximately 24 months
  MoCA is a rater-administered, participant completed assessment (PerfO instrument) used to detect cognitive impairment. It contains a series of basic assessments, including attention and visuospatial tasks. The total score ranges from 0 to 30, where lower scores indicate greater impairment.
Part 2: Number of Participants With AEs | Up to approximately 38 months
Part 2: Change From Baseline in Neurological Assessment | Up to approximately 38 months
  A neurologic examination including fundoscopy, will be performed by a neurologist or an ophthalmologist depending on local practice. A neurologic examination will include an assessment of mental status, level of consciousness, cranial nerve function, motor function, sensory function, reflexes, gait, and coordination.
Part 2: Number of Participants With Suicidal Ideation or Behavior, as Assessed by C-SSRS Score | Up to approximately 38 months
  C-SSRS measures 4 constructs as follows: severity of ideation, intensity of ideation, behavior, and lethality of actual suicide attempts. Binary (yes/no) data are collected for 10 categories. Numeric ratings are provided for intensity of ideation (if present), from 1 to 5, with 1 being the least severe and 5 being the most severe.
Part 2: Change from Baseline in MoCA | Up to approximately 38 months
  MoCA is a rater-administered, participant completed assessment (PerfO instrument) used to detect cognitive impairment. It contains a series of basic assessments, including attention and visuospatial tasks. The total score ranges from 0 to 30, where lower scores indicate greater impairment.

SECONDARY OUTCOMES:
Part 1: Plasma Concentration of RG6496 | Up to approximately 24 months
Part 1 and Part 2: Number of Participants With Anti-drug Antibody (ADA) in Plasma to RG6496 | Part 1: Up to approximately 24 months; Part 2: Up to approximately 38 months
Part 1 and Part 2: Change From Baseline of Mutant Huntingtin Protein (mHTT) Concentrations in Cerebrospinal Fluid (CSF) Over Time | Part 1: Up to approximately 24 months; Part 2: Up to approximately 38 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Westmead Hospital, Westmead, New South Wales, Australia
- New Zealand Brain Research Institute, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No